CLINICAL TRIAL: NCT02629562
Title: Single-dose, Randomised, Double-blind, Two-stage, Two-way Crossover Pharmacokinetic and Pharmacodynamic Evaluation of a Biosimilar Pegfilgrastim (B12019) Versus the Reference Product Neulasta® in Healthy Subjects
Brief Title: Pharmacokinetic and Pharmacodynamics of B12019 and Neulasta® in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cinfa Biotech (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: B12019-101
Record Dates: First submitted 2015-12-10; First posted 2015-12-14 (Estimated); Last update posted 2017-10-13 (Actual); Status verified 2016-07

CONDITIONS: Clinical Pharmacology
MeSH Terms: interventions — pegfilgrastim

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Experimental): first dosing: single dose of 6mg of B12019 administered subcutaneously, second dosing: single dose of 6mg of Neulasta administered subcutaneously
  Interventions: Biological: B12019 and Neulasta
- Arm 2 (Experimental): first dosing: single dose of 6mg of Neulasta administered subcutaneously, second dosing: single dose of 6mg of B12019 administered subcutaneously
  Interventions: Biological: B12019 and Neulasta

INTERVENTIONS:
Biological: B12019 and Neulasta — GCSF, Growth Colony Stimulating Factor

SUMMARY:
Multi-centre, double-blind, randomised, 2-way cross-over study to investigate the PK and PD of B12019 as compared to Neulasta® administered as a single subcutaneous (s.c.) dose in healthy male subjects. B12019 or Neulasta will be administered by s.c. injection.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects
* Age ≥18 and ≤55 years
* BMI 22.0 - 28.0 kg/m2
* Non-smokers for at least 6 months prior to study start
* General good health, based on a comprehensive medical history and physical examination
* Adequate organ function and normal laboratory values (unless the investigator considers an abnormality to be clinically not relevant)
* Negative hepatitis B surface antigen (HBsAg), hepatitis C antibody and human immunodeficiency virus (HIV) tests at screening
* Signed informed consent

Exclusion Criteria:

* Known hypersensitivity to Escherichia coli derived proteins, pegfilgrastim, filgrastim or any other component of B12019 or Neulasta®
* Previous exposure to filgrastim or pegfilgrastim
* History of drug or alcohol abuse
* Blood donations in the past 3 months prior to study start, or bone marrow or stem cell donor in the past 12 months (first dose)
* Medical history of haematological disease, including sickle cell disorders
* Recent infection (within 1 week prior to first dose)
* Relevant history of renal, hepatic, gastrointestinal, cardiovascular, respiratory, skin, haematological, endocrine, inflammatory or neurological diseases, that in the opinion of the investigator may interfere with the aim of the study
* Participation in an interventional or Phase I study in the last 3 months or is current a follow-up visit schedule for any study, or has participation in more than three studies of experimental drug products in the past 12 months prior to screening
* Subjects with ANC values outside the normal laboratory range at screening
* Use of prescription or over-the-counter drugs including vitamins within 4 weeks of first dosing
* Abnormalities in ECG
* Signs of dermatitis or skin abnormalities affecting the administration area and surroundings
* History of cancer

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 172 (Actual)
Dates: Start 2015-11; Primary Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
PK parameter AUC0-last | 6 weeks
  Area under the plasma concentration-time curve
PK parameter Cmax | 6 weeks
  Maximum observed drug concentration
PD parameter ANC | 6 weeks
  AUEC0-last

CONTACTS AND LOCATIONS:
Overall Officials: Michael Lissy, MD, Principal Investigator — Nuvisan GmbH
Locations (1):
- Nuvisan GmbH, Neu-Ulm, Germany